CLINICAL TRIAL: NCT03868345
Title: Speech Analysis in ALS Patients With and Without Cognitive Abnormalities: Evaluation of Sensitivity and Disease Progression
Brief Title: Speech Analysis in ALS Patients
Status: Completed | Type: Observational
Sponsor: Barrow Neurological Institute (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Jeremy Shefner, Senior Vice President and Chair of Neurology, Barrow Neurological Institute
Other Study IDs: BNI-ALS-003
Record Dates: First submitted 2019-02-06; First posted 2019-03-11 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis; Lou Gehrig Disease
Keywords: ALS; Cognitive dysfunction; Speech
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Cognitive Dysfunction; Speech

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum and blood plasma to be collected at three timepoints and retained in a biorepository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to find out if changes in speech can signal changes in the ability to think or remember. ALS patients with and without cognitive dysfunction will be followed for one year. Every three months, patients will undergo a series of cognitive and basic clinical outcomes tests. In addition, participants will take home a study-provided tablet on which they will complete weekly speech recording activities.

DETAILED DESCRIPTION:
Cognitive dysfunction is increasingly recognized as a core feature of amyotrophic lateral sclerosis (ALS). With appropriate testing, up to 50% of ALS patients will show evidence of frontotemporal dysfunction. Approximately 15% of patients meet formal criteria for frontotemporal dementia (FTD). Certain genetic forms of ALS (e.g., mutations in C9orf72) have even higher incidences of FTD. The presence of cognitive abnormalities is an adverse risk factor for survival, and its presence influences the ability of patients to cooperate in clinical trials. However, screening for frontotemporal abnormalities is frequently not performed in ALS clinics, and tools for diagnosing cognitive dysfunction are either time consuming or insensitive. Additionally, the frequently co-existing dysarthria complicates the assessment and may mask more subtle cognitive deficits. Once identified, ways of following progressive decline are also lacking. In an ongoing study, it has been shown that a sophisticated suite of speech and language analytics, developed by two of the investigators, can identify abnormalities in cognitively normal ALS patients without speech symptoms, and predict important functional changes outside of the speech domain. In this study, investigators will evaluate both speech and language in 50 patients with ALS both with and without symptoms of cognitive decline. This evaluation will be paired with two cognitive screening tools frequently used in ALS clinics, the ALS Cognitive Behavioral Screen (ALS-CBS) and the Montreal Cognitive Assessment (MoCA). The investigators will evaluate the extent to which speech and language deficits precede abnormalities as measured by the above tools and determine whether cognitive change can be accurately followed over 12 months using speech and language measures. It is hypothesized that speech and language measures will accurately and sensitively predict cognitive changes. If so, such measures may be very useful in future studies of potential therapeutic agents for ALS-FTD and other dementias.

ELIGIBILITY:
Inclusion Criteria:

1. male or female, age 21 or older,
2. diagnosed with definite, probable, or possible ALS according to the modified El Escorial Criteria,
3. a score of 2 or greater on the speech question of the ALSFRS-R (i.e. speech is intelligible with occasional repetition),
4. continuous internet access at home,
5. willingness and medical ability to comply with scheduled visits and study procedures,
6. ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations,
7. geographic accessibility to study site,
8. for the 25 participants in Group 1, NO noted symptoms of frontotemporal cognitive dysfunction, and
9. for the 25 participants in Group 2, MUST have cognitive symptoms as noted either by themselves or a caregiver.

Exclusion Criteria:

1. unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the participant's ability to comply with the protocol, and
2. any other reasons that, in the opinion of the PI, cause the candidate to be deemed unsuitable for entry into the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALS, diagnosed as definite, probable, or possible ALS according to the modified El Escorial Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in ability on Speech and Language Battery | Weekly recordings for one year
  Speech recordings made at home via a tablet using the " SpeechAssess" app.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment | Administered every three months for a year
  Cognitive screening tool
Change in ALS Cognitive Behavioral Screen | Administered every three months for a year
  Cognitive screening tool
Change in Vital Capacity | Administered every three months for a year
  Measure of breathing function
Change in Negative Inspiratory Force | Administered every three months for a year
  Measure of nasal inhale capabilities
Change in "ALS Functional Rating Scale- Revised" | Administered every three months for a year
  Questionnaire regarding daily functioning. Scale is measured from 0 to 48 points, with 48 being normal function and 0 indicating no functional abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No